CLINICAL TRIAL: NCT05702385
Title: Establishing Clinical Utility Evidence to Support Coverage and Reimbursement for Biological Dynamic's Exo-PDAC Test: A CPV® Randomized Controlled Trial
Brief Title: Clinical Utility Study for Exo-PDAC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study sponsor did not wish to proceed with the study
Sponsor: Qure Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00068105
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will enroll oncologists, interventional gastroenterologists, and primary care providers practicing in the US. Participants are randomly assigned to either control, intervention 1, or intervention 2 arms upon enrollment. All eligible and consented participants will complete two rounds of three patient simulations.
  Intervention 1 and intervention 2 arms only will receive educational material about the diagnostic test in between these two rounds. Intervention 1 arm participants only will receive the test results whether they select it or not, and Intervention 2 participants will receive the test results only if they select it in the second round of simulated cases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Practice (No Intervention): The control group treats their simulated patients using standard practice and has no introduction to the new diagnostic test.
- Intervention Group 1 - Test Results Given (Experimental): Intervention Group 1 will receive information regarding the test and will be given the test results, whether selected or not, in Round 2 of CPV administration.
  Interventions: Other: Educational Materials for a new diagnostic test
- Intervention Group 2 - Test Results Optional (Experimental): Intervention Group 2 will receive information regarding the test and will be given the test results if selected in Round 2 of CPV administration.
  Interventions: Other: Educational Materials for a new diagnostic test

INTERVENTIONS:
Other: Educational Materials for a new diagnostic test — These materials detail what the test does, how it is used, the validity and specifications of the test, and how to read its test report.
  Arms: Intervention Group 1 - Test Results Given; Intervention Group 2 - Test Results Optional

SUMMARY:
This is a national-level research study of oncologists, interventional gastroenterologists, and primary care providers. The purpose of this study is to assess the clinical evaluation and management (drug, procedures, counseling and other) of a subset of common patient care indications.

DETAILED DESCRIPTION:
The results of this study could contribute to improved quality of care for patients by encouraging better care practices and adherence to evidence-based guidance. The data from this study will be submitted to a national journal for publication. The study plans to enroll up to 250 physicians.

Upon consenting and agreeing to participate in this study, participants will be asked to care for 3 simulated patient cases, known as Clinical Performance and Value Vignettes (CPV®). CPV®s describe patients physicians typically encounter in their daily practice and are not meant to be difficult. In each vignette, physicians are asked to share their expected care through 5 domains: 1) history, 2) physical exam, 3) diagnostic workup, 4) diagnosis and 5) treatment and follow-up. Each case takes approximately 15-20 minutes to complete and we estimate the time commitment for each round of CPV® administration to be approximately 45 - 60 minutes. All responses to the cases will be completed online and will be kept confidential. Over 2 CPV® administration rounds, the total time to care for the simulated patients is estimated at 1.5-2 hours.

If physicians are randomized to an intervention group in this study, they will receive educational materials on a novel diagnostic test after the first round of CPV® administration. They are asked to review these materials before moving to the next CPV® administration round. The time to review educational materials is estimated to be approximately 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified for at least two years
* Averaging at least 20 hours per week of clinical and patient care duties over the last six months
* Routinely evaluate patients at risk for pancreatic cancer in their practice
* Practicing in the U.S.
* English speaking
* Access to the internet
* Informed, signed, and voluntarily consented to be in the study

Exclusion Criteria:

* Non-English speaking
* Unable to access the internet
* Not practicing in the U.S.
* Not averaging at least 20 hours per week of clinical or patient care duties over the last six months
* Previous exposure to the test
* Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Performance and Value (CPV)-measured variation in Assessment | [4 months]
  Measure variation in the number and quality of clinical decisions among practicing oncologists, primary care physicians, and interventional gastroenterologists in the assessment, surveillance, and management of patients at high risk of developing PDAC. The number and quality of clinical decisions will be measured on a scale of 0-100 where higher numbers represent closer adherence to evidence base national guidelines.
CPV-measured change in treatment Quality | [4 months]
  Measure of the difference in quality of overall diagnostic scores between control physicians using standard of care diagnostic tools and intervention physicians using the diagnostic test.
CPV-measured variation in evidence based decisions between control and intervention arms | [4 months]
  Measure of the difference in number of evidence-based decisions made by intervention physicians versus control physicians, while controlling for physician and practice characteristics, between rounds 1 and 2.
CPV-measured variation in evidence based decisions between intervention arms | [4 months]
  Measure the differences in amount of evidence-based decisions made by intervention group one physicians versus intervention group two physicians to assess whether the choice to order the test impacts the overall patient care and outcomes.
CPV-measured rate of adoption for the diagnostic test | [4 months]
  Rate of adoption of the test after receiving educational materials on the benefits of testing in patients who are at risk.
CPV-measured differences in cost of care between control and intervention arms | [4 months]
  Difference in the cost of care between control and intervention physicians (Cost will be calculated by measuring differential rates of medical interventions/levels of care selected by each arm, and multiplying by Medicare reimbursement rates for these interventions, and/or by modeling the incidence of expected complications and calculating associated costs per above).

CONTACTS AND LOCATIONS:
Locations (1):
- QURE Healthcare, San Francisco, California, United States